CLINICAL TRIAL: NCT01650428
Title: A Phase II, Multicentre, Open-Label, Randomised Study of Neoadjuvant Chemotherapy and Bevacizumab in Patients With MRI Defined High-Risk Cancer of the Rectum
Brief Title: Bevacizumab And Combination Chemotherapy in Rectal Cancer Until Surgery
Acronym: BACCHUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/09/0176
Record Dates: First submitted 2012-07-16; First posted 2012-07-26 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2018-10

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Bevacizumab; Neoadjuvant; Chemotherapy; Randomised
MeSH Terms: conditions — Rectal Neoplasms | interventions — Bevacizumab; Irinotecan; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFOX & Bevacizumab (Experimental): Bevacizumab - 5 mg/kg IV over 30-90 minutes (cycles 1-5 only), Oxaliplatin - 85 mg/m2 IV over 2 hours, Folinic acid - 350 mg IV over 2 hours, 5-Fluorouracil - 3200 mg/m2 IV continuous infusion over 48 hour.
  Treatment given every 2 weeks for 12 weeks (for 6 cycles)
  Interventions: Biological: Bevacizumab; Drug: Oxaliplatin; Drug: 5-Fluorouracil
- FOLFOXIRI & Bevacizumab (Experimental): Bevacizumab - 5 mg/kg IV over 30-90 minutes (cycles 1-5 only), Irinotecan - 165 mg/m2 IV over 1 hour, Oxaliplatin - 85 mg/m2 IV over 2 hours, Folinic acid - 350 mg IV over 2 hours, 5-Fluorouracil - 3200 mg/m2 IV continuous infusion over 48 hour.
  Treatment given every 2 weeks for 12 weeks (for 6 cycles)
  Interventions: Biological: Bevacizumab; Drug: Irinotecan; Drug: Oxaliplatin; Drug: 5-Fluorouracil

INTERVENTIONS:
Biological: Bevacizumab — 5 mg/kg, IV (in the vein) over 30-90 minutes, on day 1 of each 2 weekly cycles. Number of cycles: 1-5 (bevacizumab should not be administered during cycle 6).
  Other Names: Avastin
Drug: Irinotecan — 165 mg/m2 IV (intravenous) over 1 hour on day 1 of two weekly cycle. Number of cycles: 1-6
  Other Names: Campto
  Arms: FOLFOXIRI & Bevacizumab
Drug: Oxaliplatin — 165 mg/m2 IV (intravenous) over 1 hour on day 1 of two weekly cycle. Number of cycles: 1-6
  Other Names: Eloxatin
Drug: 5-Fluorouracil — 3200 mg/m2 IV (intravenous), continuous infusion over 48 hours starting on day 1 of two weekly cycle. Number of cycles: 1-6
  Other Names: 5-FU

SUMMARY:
The purpose of this study is to evaluate the efficacy, toxicity and feasibility of FOLFOX/ bevacizumab and FOLFOXIRI/ bevacizumab neoadjuvant therapy in poor prognosis rectal cancer as defined by MRI.

DETAILED DESCRIPTION:
The purpose of this study is to look at two different combinations of anticancer drugs to see how effective they are at shrinking your cancer and preventing it from coming back after surgery. Patients with locally advanced rectal cancer are sometimes treated with radiotherapy, with or without chemotherapy, before having surgery. Radiotherapy treats only the main tumour in the rectum. This means that if tiny deposits of cancer have spread to other parts of the body (metastases), these could continue to grow. Giving chemotherapy and radiotherapy together (chemoradiotherapy) can treat both the main tumour and any spread. However, due to the side-effects we can't give as much chemotherapy in combination with radiotherapy than if chemotherapy were given on its own and treatment of possible metastases may not be as good as it could be. If the risk of the main tumour coming back is quite small, then giving treatment that targets metastases should be the best option.

This study looks at two well known combinations of chemotherapy drugs: FOLFOX (folinic acid, 5-fluorouracil, oxaliplatin) and FOLFOXIRI (folinic acid, 5-fluorouracil, oxaliplatin, irinotecan). Chemotherapy works by killing cancer cells. In addition, the anticancer drug bevacizumab will be given with both the FOLFOX and FOLFOXIRI. Bevacizumab is an "anti-angiogenesis" drug. It works by stopping tumours from making new blood vessels. Without new blood vessels, the cancer cells do not get the food and oxygen they need to survive and grow. Attacking the cancer in these ways may be more effective than chemotherapy alone.

ELIGIBILITY:
Inclusion

* Histologically confirmed diagnosis of adenocarcinoma of the rectum
* Distal part of the tumour within 4-12 cm of the anal verge
* No unequivocal evidence of established metastatic disease (on chest/abdominal/pelvis CT).Patients with equivocal lesions (as determined at MDT) are eligible
* MRI-evaluated locally advanced tumour with the following:
* T3 tumours extending (≥ 4 mm), beyond the muscularis propria N0-N2
* Or tumours (involving or threatening the peritoneal surface)
* OR presence of macroscopic extramural venous invasion (V2 disease)
* AND for tumours below the peritoneal reflection, the primary tumour or involved lymph node (on MRI) must be >1 mm from the mesorectal fascia
* Measurable disease (using RECIST criteria v1.1)
* WHO performance status 0 - 1
* In the opinion of the investigator:

  * General condition considered suitable for radical pelvic surgery
  * Candidate for systemic therapy with FOLFOX/FOLFOXIRI plus bevacizumab
* Adequate bone marrow, hepatic and renal function:

  * Haemoglobin ≥80 g/L
  * ANC ≥2 x 109/L
  * Platelet count ≥100 x 109/L
  * ALT or AST ≤1.5 x ULN (upper limit of normal)
  * ALP ≤1.5 x ULN
  * Total bilirubin ≤1.5 x ULN
  * Serum creatinine ≤1.5 x ULN
  * Creatinine clearance ≥50 mL/min using the Cockcroft-Gault formula
* INR ≤ 1.1
* Urine protein ≤1+ with dipstick or urine analysis

  - For proteinuria ≥2+ or urine protein/creatinine ratio ≥ 1.0, 24-h urine protein should be obtained and the level must be ≤2 g for eligibility
* No evidence of established or acute ischaemic heart disease on ECG and normal clinical cardiovascular assessment
* No known significant impairment of intestinal absorption
* At least 18 years of age, but not more than 75 years
* Willing and able to give informed consent, comply with treatment and follow up schedule

Exclusion

* Disease outside of the mesorectal envelope (internal iliac/lateral pelvic lymph node)
* Clinically significant cardiovascular or coronary disease <2 years before randomisation
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan
* History of an arterial thromboembolic event during the previous 2 years
* Evidence of bleeding problems or coagulopathy
* Significant and continuing rectal bleeding leading to a haemoglobin <8 g/dL
* Patients receiving warfarin/coumarin derived anticoagulants at full therapeutic doses are excluded, but prophylactic doses of 1mg to prevent Hickman line clotting are eligible
* Chronic use of aspirin (>325 mg/day) or clopidogrel (>75 mg/day) within 10 days of first planned study treatment
* Require regular use of anti-diarrhoeal (e.g. daily use of loperamide)
* Serious uncontrolled intercurrent illness including poorly controlled diabetes mellitus
* Known hypersensitivity to any of the study drugs
* Serious wound, ulcer or bone fracture
* Current or impending rectal obstruction
* Metallic colonic or rectal stent in situ
* Previous pelvic radiotherapy
* Previous intolerance to fluoropyrimidine chemotherapy
* Previous treatment with bisphosphonates
* Infectious illness requiring antibiotics within 1 week of randomisation
* Previous treatment with another investigational agent within 30 days prior to randomisation
* Patients with a history of previous malignancy in the past 5 years, excepting basocellular or squamous cell skin cancer, or properly treated cervicouterine cancer in situ
* Known HIV, HBV or HCV infection
* Current smoker, or clinically relevant history of drug or alcohol abuse
* Pregnant or lactating women or pre menopausal women not using adequate contraception. Men and women of child-bearing potential must use adequate contraception
* Patients with any other condition or concurrent medical or psychiatric disease who, in the opinion of the investigator, is not eligible to enter the study
* Inability or unwillingness to comply with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2018-01-10 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response (PCR) | The pCR rate will be assessed after surgery, therefore approximately 24 weeks after randomisation.
  The proportion of patients in each arm who achieve a pCR will be presented, along with a 95% CI. Within each group the achieved pCR rate will be compared to the rate achieved by radiotherapy alone (5%).

SECONDARY OUTCOMES:
RECIST Response Rate | This will be assessed after chemotherapy has ended. Chemotherapy will be given for up to 12 weeks.
  Complete response and Partial response will be considered as responses.
CRM Negative Resection Rate | This will be assessed after surgery, therefore approximately 24 weeks after randomisation.
  Those with a resection distance >1mm amongst those having surgery.
T and N stage downstaging | This will be assessed at the completion of treatment. Treatment will be given for up to 12 weeks.
  This will examine T and N stage to assess whether stage has worsened from baseline to post-treatment. A patient will be considered to have downstaged if i) both T and N stage decrease; ii) either T or N stage decreases and the other remains stable.
Progression Free Survival | This will be assessed pre-cycle 4 and post-treatment, therefore at 6 weeks and 12 weeks after randomisation.
  This is defined as time from randomisation to disease progression or death, whichever occurs first. Disease progression will be assessed by the RECIST criteria at pre-cycle 4 and post-treatment.
Disease Free Survival | This will be length of time from date of surgery till relapse, second colorectal primary or death from any cause, whichever occurs first. These occurrences will be reported on CRFs every six months for up to three years.
  This is defined as the time from surgery with complete resections (R0) to the occurrence of relapse, second colorectal primary or death from any cause, whichever occurs first. Only subjects who have a complete resection (R0) will be included in this analysis. Patients who are alive, without recurrence and with no secondary colorectal cancer at the time of cut-off will be right-censored at the most recent date of assessment.
Overall Survival | From study entry until death, until 3 years after randomisation.
  This is defined as the time from study entry until death. The OS of all subjects and of the subgroup who had complete resection (R0) will be calculated.
Local Control | From date of surgery until local failure, until 3 years after randomisation.
  This will be assessed just for those patients who attain a CRM negative resection.
1 year Colostomy Rate | Post surgery (approximately 24 weeks after randomisation) and 1 year after randomisation.
  This will be assessed post-surgery. The Kaplan-Meier estimate will be used to estimate the colostomy rate at 1 year.
Frequency and severity of Adverse Events | This will be from date of randomisation until 30 days after completion of treatment. Treatment is given for up to 12 weeks.
  This will be tabulated for both treatment arms, including all grade 1-5 toxicities.
Compliance of Chemotherapy | This will be at the end of treatment (up to 12 weeks)
  Dose reductions and dose delays to all chemotherapy agents will be recorded.
Tumour Regression Grade (TRG) | Assessed after surgery, approximately 24 weeks after randomisation.
  This results from post-resection tumour sample will be used to categorise TRG into five groups using Dworak method.
Tumour Cell Density | This will be assessed after surgery, approximately 24 weeks after randomisation.
  This results from post-resection tumour sample will be used to provide an estimate of the average TCD and its 95% CI. This may be expressed as a mean, or if the date is skewed, the median.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Glynne-Jones, BA MB FRCP FRCR, Principal Investigator — Mount Vernon Hospital
Locations (11):
- United Kingdom (11):
  - Blackpool Victoria Hospital, Blackpool
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Charing Cross Hospital, London
  - Guy's and St Thomas' Hospital, London
  - Hammersmith Hospital, London
  - North MiddlesexHospital, London
  - Royal Marsden Hospitals NHS Foundation Trust, London
  - UCLH, London
  - Mount Vernon Hospital, Middlesex
  - Wexham Park Hospital, Slough
  - Lister Hospital, Stevenage

REFERENCES:
- [Derived] Glynne-Jones R, Hava N, Goh V, Bosompem S, Bridgewater J, Chau I, Gaya A, Wasan H, Moran B, Melcher L, MacDonald A, Osborne M, Beare S, Jitlal M, Lopes A, Hall M, West N, Quirke P, Wong WL, Harrison M; Bacchus investigators. Bevacizumab and Combination Chemotherapy in rectal cancer Until Surgery (BACCHUS): a phase II, multicentre, open-label, randomised study of neoadjuvant chemotherapy alone in patients with high-risk cancer of the rectum. BMC Cancer. 2015 Oct 23;15:764. doi: 10.1186/s12885-015-1764-1. PMID 26493588